CLINICAL TRIAL: NCT06781216
Title: Effect of Motivational Interviewing on Posttraumatic Stress Symptoms and Posttraumatic Growth in Women with Endometrial Cancer: a Randomized Controlled Trial
Brief Title: Effect of Motivational Interviewing on Posttraumatic Stress Symptoms and Posttraumatic Growth in Women with Endometrial Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Merve Kochan Aksoy, Research Assistant in Akdeniz University, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AkdenizzUniversityy
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Endometrium Cancer; Post Traumatic Stress Symptoms; Post Traumatic Growth, Psychological
Keywords: Endometrium cancer; Motivational interviewing; Post traumatic growth; Post traumatic stress symptoms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: There are two groups with parallel characteristics. The first group is the intervention group, which will be given motivational interviews. The second group is the control group without intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- motivational interviewing (Experimental): intervention group that received motivational interviewing intervention
  Interventions: Behavioral: Motivational interviewing
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: Motivational interviewing — It is emphasized that motivational interviewing is a feasible intervention that can be used by various health professionals to optimize clinical outcomes in cancer patients and survivors, helping individuals to better cope with the stress they experience related to cancer and improve their quality of life. Considering the benefits of motivational interviewing on individuals diagnosed with cancer, it is anticipated that the intervention planned in the study will improve coping strategies, reduce post-traumatic stress symptoms, and increase the level of post-traumatic growth in women with endometrial cancer.
  Arms: motivational interviewing

SUMMARY:
Cancer is still the second leading cause of death worldwide with approximately 9.6 million deaths per year. Gynecological cancers, which are the most common type of cancer among women, significantly affect the quality of life by disrupting the functions of the reproductive system of women. Endometrial cancer has an important place due to its prevalence in our country and worldwide. Although stress factors related to endometrial cancer may continue after the completion of treatment, this situation has the potential to negatively affect the psychological and physiological health of women. This research is a randomized controlled trial aiming to evaluate the effect of motivational interviewing applied to women who completed endometrial cancer treatment and were followed up in the outpatient clinic on post-traumatic stress symptoms and post-traumatic growth. Simple randomization method will be used in the study. The sample size to be included in the study was determined as 66 participants in total, 33 in the intervention group and 33 in the control group. In the study, the effectiveness of motivational interviewing technique application in women with endometrial cancer will be evaluated based on evidence using Post-Traumatic Stress Disorder Checklist for DSM-5, Post-Traumatic Growth Scale and Ways of Coping Scale. Research data will be collected from women who meet the inclusion criteria at Akdeniz University Hospital Gynecology and Obstetrics Clinic between January 2 and August 31, 2025. The motivational interviews planned to be implemented as an intervention method in the research aim to reduce post-traumatic stress symptoms, develop coping strategies and increase the level of post-traumatic growth in women with endometrial cancer.

DETAILED DESCRIPTION:
The incidence of endometrial cancer has increased in recent years, posing a serious threat to women's health, and tends to develop at a younger age. Following endometrial cancer treatment, women traditionally have regular follow-up appointments at hospital outpatient clinics to detect recurrence at an early stage, thus improving survival and support. The transition from cancer diagnosis and treatment to a long-term, rigorous surveillance protocol is a significant source of stress for individuals. Evidence suggests that endometrial cancer survivors have long-term physical, psychological, and social needs that are not met through traditional hospital-based follow-up. Previous studies have shown that the prevalence of anxiety, depression, and psychological distress in women with endometrial cancer is as high as 43.7%, 43.9%, and 54%, respectively.

Providing holistic well-being for women with endometrial cancer requires comprehensive medical, psychological, and social support throughout the course of diagnosis. As with all cancers, women with endometrial cancer who transition from primary acute treatment to follow-up survivorship face a number of significant challenges in regaining and maintaining their health and well-being. Many lack knowledge about the risk of recurrence, long-term late side effects, and how to manage them. A study of women with endometrial cancer in Australia found that women's long-term unmet needs were largely related to their psychosocial well-being, requiring assistance to cope with the expectations of themselves or others several years after their diagnosis.

When cancer becomes a part of life, individuals may experience symptoms of post-traumatic stress and even post-traumatic stress disorder. The coping mechanisms an individual uses significantly affect both psychosocial adjustment to a cancer diagnosis and play a significant role in PTG. The use of maladaptive coping strategies has also been reported to be associated with higher levels of perceived stress.

Recognizing the role of psychosocial factors in contributing to poor health outcomes and understanding individuals' coping experiences, health beliefs, and motivational factors will help design effective interventions. It is stated that motivational interviewing may be important for individuals struggling with the physical and emotional difficulties of cancer treatment or survivorship. A systematic review and meta-analysis reported that motivational interviewing has a positive effect on various health outcomes including depression and self-efficacy in the cancer population. In addition, considering the obstacles and health difficulties that these individuals face as a result of diagnosis and treatment, the study emphasizes that motivational interviewing is a feasible intervention that can be used by various health professionals to optimize clinical outcomes in cancer patients and survivors, and helps individuals better cope with the stress they experience related to cancer and improve their quality of life. Considering the benefits of motivational interviewing on individuals diagnosed with cancer, it is predicted that the intervention planned in the study will improve coping strategies in women with endometrial cancer, reduce post-traumatic stress symptoms and increase the level of post-traumatic growth.

ELIGIBILITY:
Inclusion Criteria:

* Must be a native Turkish speaker and have no communication barriers
* Have been diagnosed with endometrial cancer
* Not be in the process of active treatment (chemotherapy, radiotherapy, hormone therapy, etc.)
* Be willing to participate in the study
* Have digital literacy.

Exclusion Criteria:

* Not having mental capacity/Having a psychotic disorder
* Being in the process of active treatment (chemotherapy, radiotherapy, hormone therapy, etc.)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 66 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-08-04 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder Checklist Scale for DSM-5 | * "through study completion, an average of 1 year"
  The Post-Traumatic Stress Disorder Checklist was developed to measure the symptoms of Post-Traumatic Stress Disorder and the degree of these symptoms according to the DSM-5 diagnostic criteria. The Turkish validity and reliability of the scale was conducted by Boysan et al. in 2017. The scale, which evaluates the severity of post-traumatic stress disorder symptoms experienced by an individual in the last month after a very stressful event, consists of 20 items. The scale is a 5-point Likert-type scale and is scored as not at all = 0, very little = 1, moderately = 2, quite a lot = 3 and extremely = 4. The scores obtained from the scale range from 0 to 80, and increasing scores indicate increasing post-traumatic stress disorder symptom severity. Permission was received from the corresponding author to use the scale in research. Permission was received from the corresponding author to use the scale in research.
Post-Traumatic Growth Scale | "through study completion, an average of 1 year"
  The Posttraumatic Growth Scale was developed by Tedeschi and Calhoun in 1996 and revised in 2017. The revised Turkish version of the scale was adapted to cancer patients by Aydın and Kabukcuoğlu (2020). The scale consists of 23 items and five factors. The factors are spiritual and existential change, change in life and self-perception, personal power, new opportunities, and relationships with others. The items are scored on a 6-point Likert-type scale ranging from 0 = never experienced to 5 = experienced a lot, with higher scores indicating greater posttraumatic growth. The lowest score that can be obtained from the scale is 0 and the highest score is 115. The overall Cronbach's α of the scale was calculated as 0.93. The scale was determined to be a reliable and valid tool for Turkish cancer patient. Permission was obtained from the relevant author to use the scale in the research.
Ways of Coping Scale | "through study completion, an average of 1 year"
  The coping strategies scale was first developed by Folkman and Lazarus in 1980 with 66 items and revised in 1985. In Turkey, the 74-item version was first used by Siva (1991) by adding culturally appropriate items. The Cronbach alpha validity of the scale is .88. The scale aims to evaluate the cognitive and behavioral coping processes used by individuals after a stressful life event. The scale consists of 8 subscales: problem-focused, seeking social support, keeping a distance, delusions, self-isolation, self-blame, positivity, and stress reduction. Scale questions are rated with a four-point measurement as (0) never (3) always. Karancı et al. (1999) used this scale in their study with Dinar earthquake survivors and shortened the scale to 42 items. A total of 32 questions were removed from the scale to create a new form with 42 items, and the quadruple measurement was replaced by a triple measurement of "(0) never, (1) sometimes, (2) always". Cronbach's alpha value was found to be .76

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No